CLINICAL TRIAL: NCT01925222
Title: Effects of Pneumococcal Vaccine on Nasopharyngeal Carriage: a FinIP Effectiveness Trial Satellite Study During PCV National Vaccination Programme
Brief Title: Effects of Pneumococcal Vaccine on Nasopharyngeal Carriage
Status: Completed | Type: Observational
Sponsor: Arto Palmu (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Arto Palmu, Research manager, Finnish Institute for Health and Welfare
Organization: Finnish Institute for Health and Welfare (Other Government)
Other Study IDs: FinIP-carriage13THL
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Nasopharyngeal Carriage of Streptococcus Pneumoniae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasopharyngeal and oropharyngeal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- PCV-vaccinated infant, 3+1 schedule
- PCV-vaccinated infant, 2+1 schedule
- Control-vaccinated infant
- PCV-vaccinated child, catch-up schedule
- Control-vaccinated child, catch-up schedule

SUMMARY:
The purpose of this study is to assess the direct effects of the ten-valent pneumococcal conjugate vaccine administered to infants on nasopharyngeal carriage at 3 to 5 years of age.

These children have been vaccinated in infancy in the cluster-randomized Finnish Invasive pneumococcal Disease (FinIP) Trial (a separate protocol reported at ClinicalTrials.gov Identifier:NCT00861380) during 2009 to 2011.

Also the indirect effect on nasopharyngeal carriage will be assessed on vaccinees' elder non-vaccinated siblings aged 5 to 9 years.

DETAILED DESCRIPTION:
This study includes a cross-sectional sampling of nasopharyngeal and oropharyngeal swabs in 2013 from vaccinated and unvaccinated children.

ELIGIBILITY:
Inclusion Criteria for FinIP-vaccinated children:

1. age 3 to 5 years
2. enrolled in the FinIP trial and has received at least one dose of study vaccine in the infant vaccine schedule (3+1 or 2+1)
3. at least one parent with fluent Finnish
4. informed consent from one parent

Exclusion criteria for FinIP-vaccinated children

1. PCV vaccination administered, other than the randomized study vaccine
2. history of antimicrobial treatment within 4 weeks (the child can be enrolled later)

Inclusion criteria for unvaccinated siblings

1. age 5 to 9 years
2. younger sibling living in the same household having participated in the FinIP trial (regardless of the vaccination schedule)
3. at least one parent with fluent Finnish
4. informed consent from one parent

Exclusion criteria for unvaccinated siblings

1. PCV vaccination administered
2. history of antimicrobial treatment within 4 weeks (the child can be enrolled later)

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children vaccinated in infancy in the cluster-randomized Finnish Invasive pneumococcal Disease (FinIP) Trial (ClinicalTrials.gov Identifier:NCT00861380) during 2009 to 2011 and their unvaccinated older siblings.
Sampling Method: Non-Probability Sample
Enrollment: 3900 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Carriage due to any pneumococcal serotype included in the ten-valent pneumococcal conjugate vaccine (PCV10) in children vaccinated in infancy | one sampling at 3 to 5 years of age
  Nasopharyngeal and oropharyngeal swabs taken once at 3 to 5 years of age

SECONDARY OUTCOMES:
Carriage due to any pneumococcal serotype in children vaccinated in infancy | one sampling at 3 to 5 years of age

OTHER OUTCOMES:
Carriage due to any pneumococcal serotype included in the PCV vaccine in unvaccinated older siblings of the PCV10-vaccinated children | one sampling at 5 to 9 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Arto A Palmu, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Tampere, Finland

REFERENCES:
- [Background] Palmu AA, Jokinen J, Borys D, Nieminen H, Ruokokoski E, Siira L, Puumalainen T, Lommel P, Hezareh M, Moreira M, Schuerman L, Kilpi TM. Effectiveness of the ten-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10) against invasive pneumococcal disease: a cluster randomised trial. Lancet. 2013 Jan 19;381(9862):214-22. doi: 10.1016/S0140-6736(12)61854-6. Epub 2012 Nov 16. PMID 23158882
- See also: Public webpage for the FinIP trial and the carriage study — http://www.finip.fi